CLINICAL TRIAL: NCT00669097
Title: An Open-Label, Non-Randomized, Single-Center, Phase I Study to Determine the Absorption, Distribution, Metabolism and Excretion (ADME) of TKI258 After a Single Oral Administration of TKI258 500mg and to Assess the Preliminary Safety of TK258 400mg Once Daily in Patients With Advanced Solid Malignancies
Brief Title: Absorption, Distribution, Metabolism and Excretion (ADME) Study of TKI258 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2106
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2011-08

CONDITIONS: Advanced Solid Malignancies
Keywords: ADME; TKI258; RTKs inhibitor; PDGRF inhibitor; VEGFER inhibitor
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
This is a phase l study to examine Absorption, Distribution, Metabolism and Excretion of TKI258. There are 2 cohorts. Cohort 1 (4 patients) will receive single radio-labeled 500mg dose of TKI258 followed after 15 days by daily dosing of 400mg TKI258. Cohort 2 (9 patients) will receive 400mg TKI258.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥ 18 years
2. Patients with histologically confirmed solid tumor or lymphoma who are resistant/refractory to approved therapies or for whom no appropriate therapies are available.
3. WHO performance status ≤ 2
4. All previous treatment (including surgery and radiotherapy) must have been completed at least four weeks prior to study entry and any acute toxicities must have been resolved
5. Written informed consent to participate in the study

Exclusion criteria:

1. Primary Brain Tumors or symptomatic leptomeningeal metastases
2. Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within six months of study start
3. Fertile males not willing to use contraception or whose female partners are not using adequate contraceptive protection Pregnant or lactating women (all women of childbearing potential must have a negative pregnancy test (> 5 mIU/ml) before inclusion in the study; post-menopausal women must be amenorrheic for at least 12 months). Female patients must use adequate contraceptive protection
4. Centrally located or squamous cell carcinoma of the lung
5. Proteinuria > 1+ on dipstick testing
6. History of gastrointestinal malabsorption Surgery involving intestinal anastomosis within four weeks of study start.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Cohort1: Find out about the routes and rates of excretion of TKI258 and its metabolites | Day 15
Cohort 2: Safety and Tolerability of TKI258 | Time to patient withdrawal due to disease progression or tolerability issues

SECONDARY OUTCOMES:
Cohort 1: Safety and tolerability of TKI258 | Time to patient withdrawal due to disease progression or tolerability issues
Cohort 1: Preliminary anti-tumor activity of TKI258 | Time to tumor progression
Preliminary Anti-tumor activity of TKI258 | Time to tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Amsterdam, Netherlands

REFERENCES:
- [Derived] Dubbelman AC, Upthagrove A, Beijnen JH, Marchetti S, Tan E, Krone K, Anand S, Schellens JH. Disposition and metabolism of 14C-dovitinib (TKI258), an inhibitor of FGFR and VEGFR, after oral administration in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2012 Nov;70(5):653-63. doi: 10.1007/s00280-012-1947-2. Epub 2012 Aug 22. PMID 23010851
- See also: Results for CTKI258A2106 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4883